CLINICAL TRIAL: NCT04825574
Title: Extension Protocol for Patients Previously Treated in Avapritinib Clinical Trials
Brief Title: Study for Patients Previously Treated in Avapritinib Clinical Trials
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BLU-285-1408
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-10

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — avapritinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patients with GIST previously enrolled in avapritinib clinical trials (Experimental)
  Interventions: Drug: Avapritinib

INTERVENTIONS:
Drug: Avapritinib — avapritinib tablet
  Other Names: BLU-285

SUMMARY:
This is an open-label extension study to provide long term safety data for GIST patients who are deriving clinical benefit from avapritinib upon the completion of avapritinib clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has histologically confirmed metastatic or unresectable GIST as established by entry in a previous avapritinib clinical trial and has been receiving treatment with avapritinib on one of these trials.
2. Patient continues to receive clinical benefit from avapritinib treatment, as assessed by the investigator.
3. Patient or legal guardian, if permitted by local regulatory authorities, provides informed consent.

Exclusion Criteria:

1. Patient requires therapy with a concomitant medication that is a strong inhibitor or strong inducer of cytochrome P450 (CYP) 3A4
2. Patient has a history of intracranial bleeding either prior to or during avapritinib treatment
3. Patients who have poor organ function, defined as Adverse Events of NCI CTCAE version 5.0 Grade 3 or higher at the time of enrollment must delay start of treatment until symptoms return to Grade 2 or baseline, or the start of treatment has been approved by the Sponsor.
4. Patients who have ongoing cognitive or mood effects Adverse Events of NCI CTCAE version 5.0 higher than Grade 1 must delay start of treatment until symptoms return to Grade 1 or baseline.
5. Women who are unwilling, if not postmenopausal or surgically sterile, to abstain from sexual intercourse or employ highly effective contraception from the time of enrollment and for at least 30 days after the last dose of avapritinib. Men who are unwilling, if not surgically sterile, to abstain from sexual intercourse or employ highly effective contraception from the time of first dose and for at least 90 days after the last dose of avapritinib.
6. Women who are pregnant.
7. Women who are breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2023-11-23 (Actual); Study Completion 2023-11-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Gustave Roussy Cancer Campus Grand Paris Institut de Cancerologie Gustave-Roussy, Villejuif, Val-de-Marne, France

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two participants (one from BLU-285-1101 (NCT02508532) and one from BLU-285-1303 (NCT03465722)) were continuing to receive avapritinib and were enrolled in this extension study.
Groups:
- Avapritinib: Participants with gastrointestinal stromal tumor (GIST) who were deriving clinical benefit from avapritinib upon the completion of avapritinib clinical studies received avapritinib once daily (QD) at the specified dose of the prior avapritinib protocol.
Period: Overall Study
Arm/Group | Avapritinib
Started | 2
Received at Least 1 Dose of Study Drug | 2
Completed | 0
Not Completed | 2
Not completed — Commercial treatment became available | 1
Not completed — Disease progression | 1

BASELINE CHARACTERISTICS:
Population: The Safety Population was defined as all participants who received at least one dose of avapritinib. Baseline measure data are not reported for participant privacy reasons due to low enrollment
Groups:
- Avapritinib: Participants with GIST who were deriving clinical benefit from avapritinib upon the completion of avapritinib clinical studies received avapritinib QD at the specified dose of the prior avapritinib protocol.
Arm/Group | Avapritinib
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants] — Population: The Safety Population was defined as all participants who received at least one dose of avapritinib. Baseline measure data are not reported for participant privacy reasons due to low enrollment
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The Safety Population was defined as all participants who received at least one dose of avapritinib. Baseline measure data are not reported for participant privacy reasons due to low enrollment
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The Safety Population was defined as all participants who received at least one dose of avapritinib. Baseline measure data are not reported for participant privacy reasons due to low enrollment
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The Safety Population was defined as all participants who received at least one dose of avapritinib. Baseline measure data are not reported for participant privacy reasons due to low enrollment

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: AESIs for avapritinib are, regardless of grade or causality:
  * cognitive effects which include the following terms: memory impairment, cognitive disorder, confusional state and encephalopathy.
  * intracranial bleeding including haemorrhage intracranial, cerebral haemorrhage , and subdural haematoma.
Time Frame: From date of first avapritinib dose through 30 days after the last avapritinib dose (up to approximately 31 months)
Population: The Safety Population was defined as all participants who received at least one dose of avapritinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Avapritinib
Number analyzed (Participants) | 2
Participants | 0

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAEs were defined as death, a life-threatening AE, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event that jeopardized participant and required medical intervention to prevent 1 of the outcomes listed in this definition. A summary of all serious AEs, regardless of causality is located in Reported AE section.
Time Frame: From date of first avapritinib dose through 30 days after the last avapritinib dose (up to approximately 31 months)
Population: The Safety Population was defined as all participants who received at least one dose of avapritinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Avapritinib
Number analyzed (Participants) | 2
Participants | 1

ADVERSE EVENTS:
Time Frame: From date of first avapritinib dose through 30 days after the last avapritinib dose (up to approximately 31 months)
Description: The Safety Population was defined as all participants who received at least one dose of avapritinib. As specified in the protocol, only SAEs and AESIs were collected. Non-serious adverse event data was not collected.
Arm/Group | Avapritinib
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Avapritinib (N=2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/74/NCT04825574/Prot_SAP_000.pdf